CLINICAL TRIAL: NCT06905418
Title: Design and Validation of a Mobile Health Application for Home-Based Musculoskeletal Therapy in Ankle Sprain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/782
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic (Experimental)
  Interventions: Diagnostic Test: Clinic
- Mobile App (Experimental)
  Interventions: Combination Product: Mobile App

INTERVENTIONS:
Diagnostic Test: Clinic — group A will get treatment in clinic
  Arms: Clinic
Combination Product: Mobile App — group B will use mobile application for treatment
  Arms: Mobile App

SUMMARY:
"Ankle sprain is a common musculoskeletal injury that can pointedly influence the quality of life of an indivual. Old rehabilitation approaches often require recurrent clinic visits, which can be time-consuming, costly, and unreachable to many. This study aims to design and validate a mobile health application for home-based musculoskeletal therapy in ankle sprain.

DETAILED DESCRIPTION:
The study will employ a randomized controlled trial design, involving patients with ankle sprains, healthcare professionals, and healthy volunteers. The mobile health application will be designed to provide personalized exercises, education, and monitoring to improve rehabilitation outcomes. The study will evaluate the effects of the mobile health application (m Health) in reducing pain, improving functional ability, and ornamental quality of life. The study will also assess the usability and acceptability of the application among patients and healthcare professionals.

Outcome measurement tools will contain the Foot and Ankle Ability Measure (FAAM), Numeric Pain Rating Scale (NPRS) and System Usability Scale (SUS) The study will contribute to the development of an innovative, home-based rehabilitation solution for individuals with ankle sprains, improving accessibility and adherence to rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-65 years, both gender(male and female) will be included.
* Include participants clinically diagnosed with a lateral ankle sprain confirmed by a healthcare professional, with a clear timeframe such as within the last 4-6 weeks.
* Grade I and II sprains (mild to moderate) will be included using NPRS tool range from 0 to 6.
* Participants must own and be able to use a smartphone or tablet that is compatible with the mobile health application.
* Specify that participants must be able to read and understand the application interface language.
* Ensure participants can safely perform the exercises prescribed in the app without additional risk of injury

Exclusion Criteria:

* Concurrent fractures of the leg or foot.
* Previous surgery in the affected ankle or surgery resulting from the current ankle sprain.
* Serious systemic illnesses (e.g. rheumatoid arthritis, or fibromyalgia).
* Neurological impairments or other conditions that may affect rehabilitation outcomes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | 12 Months
  FAAM. Each item of the FAAM is scored on a 5-point Likert scale with 4 points representing no difficulty at all; 3 points, slight difficulty; 2 points, moderate difficulty; 1 point, extreme difficulty; and 0 points, unable to do
Numeric pain rating scale (NPRS) | 12 months
  The Numeric Pain Rating Scale (NPRS) is perhaps the most frequently applied scale used to quantify pain intensity in the clinical setting. It is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No